CLINICAL TRIAL: NCT03588182
Title: Virtual Reality Analgesia for External Cephalic Version
Brief Title: Virtual Reality for External Cephalic Version
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAR9073
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Analgesia Management for External Cephalic Version
Keywords: Virtual Reality (VR)

STUDY DESIGN:
Intervention Model Description: Parallel design, nonblinded, randomized controlled superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group VR (Experimental): Virtual reality (VR) experience VR visualization of a 3-dimensional relaxing nature scene with the accompanying audio. The patient will be offered a selection of scenes from which to choose, played continuously on a Samsung Gear VRTM(San Jose, CA) headset and headphones. The goal is for the patient to use the intervention for the entire duration of the external cephalic version procedure (ECV), which typically lasts 15 - 30 minutes.The patient will also receive verbal reassurance and coaching as needed. The obstetrician will communicate as usual with the patient.
  Interventions: Other: Virtual Reality Experience
- Group No VR (No Intervention): No intervention will be provided for the control group, who will receive usual management at CUMC, which involves provision of no analgesia or sedation for the procedure, which typically lasts 15 - 30 minutes. Verbal reassurance and coaching is routinely provided by caregivers, including encouraging deep breathing, particularly during painful manipulation of the abdomen, for the duration of the procedure. The obstetrician will communicate as usual with the patient - for example advising that he/she is about to begin the procedure and giving updates as to the degree of success.

INTERVENTIONS:
Other: Virtual Reality Experience — Virtual reality visualization and experience of a 3-dimensional relaxing nature scene with the accompanying audio.
  Arms: Group VR

SUMMARY:
This will be a parallel design, nonblinded, randomized controlled superiority trial investigating the utility of a virtual reality (VR) experience to provide analgesia for external cephalic version (ECV).

DETAILED DESCRIPTION:
Subjects will be: Pregnant women, age >18 years, with a singleton pregnancy at >36 weeks gestational age, healthy (American Society of Anesthesiologists physical status class II), with an otherwise uncomplicated pregnancy (i.e. no fetal abnormalities or significant maternal morbidity, scheduled for ECV at Columbia University Irving Medical Center (CUIMC) with a plan to receive no anesthesia for the procedure.

Patients will be randomly assigned to either the VR or No VR group. The intervention will be provided for the duration of the ECV procedure (typically 15 - 30 mins).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women, age >18 years, with a singleton pregnancy at >36 weeks gestational age, healthy (American Society of Anesthesiologists physical status class II), with an otherwise uncomplicated pregnancy (i.e. no fetal abnormalities or significant maternal morbidity, scheduled for ECV at CUMC with a plan to receive no anesthesia for the procedure.

Exclusion Criteria:

* 1) severe claustrophobia or other psychological/psychiatric disorder which would prevent the use of a VR headset; 2) history of severe motion sickness, which may lead to nausea and vomiting or other discomfort with use of the a VR headset; 3) severe visual impairment, which may prevent appreciation of the visual aspects of the VR environment presented; 4) severe auditory impairment, which may prevent full appreciation of the sounds presented in the VR environment; 5) facial skin or scalp open lesions which could be irritated or risk infection to the patient or others if the VR headset is used; 6) other viral/bacterial/fungal infectious illnesses that could easily be spread by sharing of the device e.g. viral or bacterial conjunctivitis, meningitis, influenza, common cold, and other upper respiratory tract infections; 7) severe or uncontrolled seizure disorder, as the VR experience could invoke seizures 8) bulky hairstyles which would significantly impair correct fitting of the VR headset.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 5 (Actual)
Dates: Start 2019-05-18 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Mean maximal numerical rating scale (NRS) score ( scale 0 - 10) for pain during the ECV procedure. | The maximal rated pain score will be determined within 5 minutes of the end of the ECV procedure.
  Verbal rating of pain (scale 0 - 10) during ECV procedure, rated every 5 minutes

SECONDARY OUTCOMES:
Success of ECV procedure | Within 5 minutes of the end of the ECV procedure
  The successful manipulation of the fetus from the breech to cephalic position
Rating of the likelihood of choosing the analgesia technique received again | Within 2 hours of the end of the procedure
  Verbal rating of likelihood to choose the analgesia technique received again (scale 1 - 5, where 1 = I would not utilize again, 5 = I would definitely utilize again)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lee, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
An excel spreadsheet with data will be available on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After data analysis, for an indefinite period of time
Access Criteria: An excel spreadsheet with data will be available on request.